CLINICAL TRIAL: NCT00336297
Title: Testing Screening Formats for Indicator-Based and Universal Screening Measurements in the Identification of Woman Abuse.
Brief Title: Testing Methods of Screening for Woman Abuse in Health Care Settings.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ontario Women's Health Council (Unknown)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MacMillan_VAW_Testing_Trial
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2005-02

CONDITIONS: Domestic Violence
Keywords: screening; screening methods; intimate partner violence

INTERVENTIONS:
Procedure: Woman Abuse Screening Tool
Procedure: Partner Violence Screen
Procedure: Computerized screening
Procedure: Face to face screening
Procedure: Written screening on forms

SUMMARY:
Recent reviews have identified the need for additional high quality exploratory and evaluative research to understand 1) the actual impact on all women of instituting mass screening procedures versus using indicator-based approaches to identifying woman abuse and 2) the extent to which early identification through screening -- either universal or indicator-based is effective in preventing or ameliorating important outcomes. This is a critical first step in developing a larger randomized controlled trial (RCT) which examines the effectiveness of screening in preventing woman abuse, improving quality of life and other associated outcomes. This study prepares for the RCT by testing the optimal method of administration for the two screening instruments that will be used in the RCT. The administration formats are: computer-based screen, paper and pencil screen and face-to-face screen. They study will also determine recruitment rates.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-64 years
* Patients at the health care site
* Able to participate in English
* Able to separate from accompanying person(s)

Exclusion Criteria:

* Too ill to participate
* Unable to separate from accompanying person(s)
* Unable to speak, read, or write English

Ages: 18 Years to 64 Years | Sex: Female
Age Groups: Adult
Enrollment: 2000
Dates: Start 2004-05; Study Completion 2005-02

PRIMARY OUTCOMES:
disclosure rates for past year exposure to intimate partner violence

SECONDARY OUTCOMES:
participant satisfaction with completing the instruments
missing data

CONTACTS AND LOCATIONS:
Overall Officials: Harriet L MacMillan, MD, MSc, Principal Investigator — McMaster University
Locations (7):
- Canada (7):
  - Cambridge Memorial Hospital - Emergency Department, Cambridge, Ontario
  - Carlisle Medical Centre, Carlisle, Ontario
  - City of Hamilton Public Health and Community Services Department, Hamilton, Ontario
  - Hamilton Health Sciences Colposcopy Clinic, Hamilton, Ontario
  - Victoria Family Medical Centre, London, Ontario
  - London Health Sciences - Victoria Hospital Clinic 5A, London, Ontario
  - Norfolk General Hospital - Emergency Department, Simcoe, Ontario

REFERENCES:
- [Result] MacMillan HL, Wathen CN, Jamieson E, Boyle M, McNutt LA, Worster A, Lent B, Webb M; McMaster Violence Against Women Research Group. Approaches to screening for intimate partner violence in health care settings: a randomized trial. JAMA. 2006 Aug 2;296(5):530-6. doi: 10.1001/jama.296.5.530. PMID 16882959
- See also: Protocol for the subsequent RCT of effectiveness of screening for intimate partner violence. — http://www.clinicaltrials.gov/ct/show/NCT00182468?order=1